CLINICAL TRIAL: NCT02852564
Title: Ethacrynic Acid Elimination in Non-Muscle Invasive Bladder Cancer Patients Undergoing Transurethral Resection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eugene Lee, MD (Other)
Collaborators: University of Kansas Medical Center (Other)
Responsible Party: Sponsor-Investigator, Eugene Lee, MD, Medical Doctor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015IITEthacrynicAcidBladderCa
Record Dates: First submitted 2016-06-28; First posted 2016-08-02 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Bladder Cancer
Keywords: Non-Muscle; Invasive; Bladder; Cancer; Muscle; Surgery; Transurethral; Resection; Tumor; Ethacrynic; Acid; Mitomycin; Urine; NMIBC
MeSH Terms: conditions — Urinary Bladder Neoplasms; Neoplasms; Heartburn; Non-Muscle Invasive Bladder Neoplasms | interventions — Ethacrynic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Enrolled Participants (Experimental): Administration of a single, 50 mg oral dose of ethacrynic acid prior to bladder tumor removal surgery (Transurethral Resection of Bladder Tumor [TURBT])
  Interventions: Drug: Ethacrynic Acid

INTERVENTIONS:
Drug: Ethacrynic Acid — One oral dose at 50 mg prior to bladder tumor removal surgery
  Other Names: Edecrin

SUMMARY:
Phase 1 study to provide quantitative characterization of the renal elimination of ethacrynic acid and metabolites in patients with non-muscle invasive bladder cancer (NMIBC) at the time of transurethral resection of bladder tumor

DETAILED DESCRIPTION:
Bladder cancer continues to be a significant healthcare and financial liability in the United States. Patients with Non-Muscle Invasive Bladder Cancer (NMIBC) are in desperate need for both effective and easily tolerated treatment options. Current standard of care includes immediate post-operative Mitomycin C (MMC), which decreases the rate of recurrence but does not alter progression. Furthermore, in patients with high-grade NMIBC, standard of care dictates that patients undergo intravesical Bacillus Calmette-Guerin (BCG) therapy. This treatment has a high degree of morbidity with both local and systemic side effects along with significant discomfort from treatment (intra-urethral catheterization and bladder instillation). Our goal is to develop a bladder cancer treatment strategy designed to decrease recurrence/progression rates in addition to decreasing the morbidity of treatment.

Twelve evaluable NMIBC patients will participate in this Phase 1 trial.

Treatment - patients will receive a single, 50 mg oral dose of ethacrynic acid administered as two 25 mg strength EDECRIN® tablets immediately prior to transurethral resection of bladder tumor.

Concentrations and excretion rates of ethacrynic acid in the urine, as well as of cysteine, glutathione, and mercapturate metabolites, will be measured for each of 4 urine specimens collected on the day of surgery (before, during, and at 2 timepoints after surgery).

Adverse events, serious adverse events, laboratory values, and vital sign measurements will be collected.

Efficacy of ethacrynic acid treatment will be estimated by recording recurrence/non-recurrence of disease at 3 months post-treatment

ELIGIBILITY:
INCLUSION CRITERIA:

NOTE: Both patients who will and will not receive standard of care concomitant mitomycin C are eligible to enroll in this study.

* Ability to understand and the willingness to sign a written informed consent
* Diagnosis of presumed non-muscle invasive bladder cancer based on office based cystoscopy (primary or recurrent), and planned transurethral resection of bladder tumor (TURBT)
* Participants must have tumors with anticipated transurethral resection time ≤ 1 hour
* Previous history of intravesical therapy allowed
* Age ≥ 18 years
* Performance Status 0-1
* Adequate organ and marrow function as defined below:

  * leukocytes ≥ 3,000/mcL
  * absolute neutrophil count ≥ 1,500/mcL
  * platelets ≥ 100,000/mcl
  * total bilirubin within normal institutional limits
  * Aspartate Aminotransferase (AST) ≤ 2.5 X institutional upper limit of normal
  * Alanine Aminotransferase (ALT) ≤ 2.5 X institutional upper limit of normal
  * creatinine ≤ 2.5 X institutional upper limit of normal
* Women of child-bearing potential (WOCP) and men with partners of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately *A woman of child-bearing potential is any female (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

  * Has not undergone a hysterectomy or bilateral oophorectomy; or
  * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months)

EXCLUSION CRITERIA:

Participants meeting any of the exclusion criteria at baseline will be excluded from study participation.

* Current or anticipated use of other investigational agents.
* Patient has known nodal or distant metastatic disease. Patients with nodal or metastatic disease require systemic chemotherapy. Furthermore, they should be excluded from this clinical trial because of their poor overall prognosis.
* Patients with locally advanced bladder cancer based on cross-sectional imaging (suspicion of extravesical disease or hydronephrosis)
* Patients with tumors with anticipated transurethral resection time greater than 1 hour
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Ethacrynic acid or other agents used in study.
* Systolic blood pressure < 90 mmHg and/or diastolic blood pressure < 50 mmHg
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or nursing. There is a potential for congenital abnormalities and for this regimen to harm nursing infants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Urine Concentration - Ethacrynic Acid and its conjugates | Baseline at 30 minutes before surgery
  Concentration of Ethacrynic acid and its conjugates in urine for baseline at 30 minutes before surgery. A: Ethacrynic acid concentration (ng/mL) B: Glutathione (ng/mL) C: Cysteine (ng/mL) D: Mercapturic acid (ng/mL) will be measured.
Urine Concentration - Ethacrynic Acid and its conjugates | During surgery
  Concentration of Ethacrynic acid and its conjugates in urine during surgery. A: Ethacrynic acid concentration (ng/mL) B: Glutathione (ng/mL) C: Cysteine (ng/mL) D: Mercapturic acid (ng/mL) will be measured.
Urine Concentration - Ethacrynic Acid and its conjugates | 2 hours after surgery
  Concentration of Ethacrynic acid and its conjugates in urine at 2 hours after surgery. A: Ethacrynic acid concentration (ng/mL) B: Glutathione (ng/mL) C: Cysteine (ng/mL) D: Mercapturic acid (ng/mL) will be measured.
Urine Concentration - Ethacrynic Acid and its conjugates | 4 hours after surgery
  Concentration of Ethacrynic acid and its conjugates in urine at 4 hours after surgery. A: Ethacrynic acid concentration (ng/mL) B: Glutathione (ng/mL) C: Cysteine (ng/mL) D: Mercapturic acid (ng/mL) will be measured.
Excretion Rates - Ethacrynic Acid and its conjugates | 30 minutes before surgery
  Urinary excretion rates of ethacrynic acid and its conjugates for baseline at 30 minutes before surgery. A: Ethacrynic acid concentration (ng) B: Glutathione (ng) C: Cysteine (ng) D: Mercapturic acid (ng) will be measured.
Excretion Rates - Ethacrynic Acid and its conjugates | during surgery
  Urinary excretion rates of ethacrynic acid and its conjugates during surgery. A: Ethacrynic acid concentration (ng) B: Glutathione (ng) C: Cysteine (ng) D: Mercapturic acid (ng) will be measured.
Excretion Rates - Ethacrynic Acid and its conjugates | 2 hours after surgery
  Urinary excretion rates of ethacrynic acid and its conjugates 2 hours after surgery.
  A: Ethacrynic acid concentration (ng) B: Glutathione (ng) C: Cysteine (ng) D: Mercapturic acid (ng) will be measured.
Excretion Rates - Ethacrynic Acid and its conjugates | 4 hours after surgery
  Urinary excretion rates of ethacrynic acid and its conjugates 4 hours after surgery.
  A: Ethacrynic acid concentration (ng) B: Glutathione (ng) C: Cysteine (ng) D: Mercapturic acid (ng) will be measured.

SECONDARY OUTCOMES:
Number of Participants with treatment-related adverse events as assessed by CTCAE 4.03 | During and after surgery, up to 3 months following surgery
  Adverse events / toxicity related to Ethacrynic Acid as reported by participants will be recorded. Toxicity will be measured via analysis of patient adverse events (physiological parameter). Adverse events will be scored using NCI Common Toxicity Criteria for Adverse Events v 4.0.3 (June 14,2010).
Number of Participants with Tumor Recurrence / Non-Recurrence using RECIST version 1.1 | 90 days after surgery
  Tumor Recurrence / Non-Recurrence will be measured using RECIST version 1.1 to assess efficacy of ethacrynic acid

CONTACTS AND LOCATIONS:
Overall Officials: Eugene K Lee, MD, Principal Investigator — The University of Kansas - Cancer Center
Locations (1):
- The University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: Undecided